CLINICAL TRIAL: NCT05245409
Title: The Relationship Between Stress Scores, a Single-session of Chiropractic Care, Heart Rate Variability, and Electroencephalography Patterns
Brief Title: Stress, EEG, ECG, and Chiropractic
Acronym: BLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: I-0016
Record Dates: First submitted 2022-01-27; First posted 2022-02-18 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Stress
Keywords: stress, chiropractic, EEG, HRV

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress (Experimental): Individuals under various degrees of stress
  Interventions: Other: Chiropractic adjustment using an activator

INTERVENTIONS:
Other: Chiropractic adjustment using an activator — Chiropractic adjustment using an activator

SUMMARY:
The Life University Center for Chiropractic Research is conducting a study to better understand the relationship between subjective stress measures and brain patterns during resting state and an auditory oddball task. A secondary aim is to evaluate the impact of a single session of chiropractic care on the resting state and P300 time locked response after a one-week wait period. An additional outcome assessment for this study will be the recording of an electrocardiogram (ECG) of each participant that will be used to analyze their heart rate variability (HRV). Eligible individuals will receive a physical exam to ensure safety during all procedures. They will then sit for a 6-minute resting state EEG and an auditory oddball task. They will complete a series of questionnaires assessing stress. They will receive a chiropractic adjustment using a handheld instrument called an Activator. They will return one week later for a follow-up assessment consisting of the 6-minute resting state EEG, auditory oddball task, and the questionnaires assessing stress.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18 and 40
* Individuals who can wear an EEG cap for 40 minutes
* Individuals who can sit quietly for at least 15 minutes
* Individuals who have not had a chiropractic adjustment within the last two weeks
* Individuals who have not received any other interventions, such as osteopathic spinal manipulation, physical therapy rehabilitation or manipulation, massage, body movement therapies or acupuncture within the last 2 weeks.

Exclusion Criteria:

* Individuals who have been diagnosed with a serious mental disorder such as schizophrenia or major depressive disorder that could influence EEG results
* Individuals who do not feel they can sit quietly with limited movement for roughly 15 minutes
* Individuals who are on psychotropic medications (e.g. Benzodiazepine medications) that influence EEG readings (Benzodiazepine medications include but are not limited to: alprazolam, chlordiazepoxide, clobazam, clonazepam, clorazepate, diazepam, estazolam, flurazepam, lorazepam, midazolam, oxazepam, temazepam, triazolam, etc.)
* Individuals with any injury or surgery to the skull in the last 6 months, or a history of trauma to the head such as a concussion or stroke
* Individuals with a hearing impairment (due to the auditory stimulus recording being performed)
* Individuals who are currently pregnant
* Individuals with a current litigation related to a physical, health-related injury
* Individuals with untreated diagnosed osteoporosis or articular instability, such as atlanto-axial instability
* Individuals with a known heart condition that results in an aberrant ECG recording

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Electroencephalography Power spectrum | Baseline (Pre)
  6 minutes of resting state EEG with eyes closed. 64 channels of EEG will be recorded. A fast Fourier transform will be computed to provide a power spectrum of frequencies 1-50.
Electroencephalography Power spectrum | one-week (post)
  6 minutes of resting state EEG with eyes closed. 64 channels of EEG will be recorded. A fast Fourier transform will be computed to provide a power spectrum of frequencies 1-50.
Auditory oddball task | Baseline (Pre)
  Auditory oddball task with 200 common and 40 rare stimuli. P300 evoked related potential evaluated through capturing EEG.
Auditory oddball task | one-week (post)
  Auditory oddball task with 200 common and 40 rare stimuli. P300 evoked related potential evaluated through capturing EEG.
Heart rate variability (HRV) | Baseline (Pre)
  ECG recording will be used to evaluate HRV from R-R intervals.
Heart rate variability (HRV) | one-week (post)
  ECG recording will be used to evaluate HRV from R-R intervals.
Weekly Stress Inventory Short Form | Baseline (Pre)
  25 questions. Likert scale: did not happen; happended but not successful; slightly stressful; mildly stressful; moderately stressful; stressful; very stressful; extremely stressful.
Weekly Stress Inventory Short Form | one-week (post)
  25 questions. Likert scale: did not happen; happended but not successful; slightly stressful; mildly stressful; moderately stressful; stressful; very stressful; extremely stressful.
Hamilton Anxiety Rating Scale | Baseline (pre)
  14 questions. Likert scale: not true at all; rarely true; sometimes true; often true; true nearly all the time.
Hamilton Anxiety Rating Scale | one-week (post)
  14 questions. Likert scale: not true at all; rarely true; sometimes true; often true; true nearly all the time.
Connor Davidson Resilience Scale - 25 | baseline (pre)
  25 questions. Likert scale: not true at all; rarely true; sometimes true; often true; true nearly all the time.
Connor Davidson Resilience Scale - 25 | one-week (post)
  25 questions. Likert scale: not true at all; rarely true; sometimes true; often true; true nearly all the time.
Severity of Acute Stress Symptoms | baseline (pre)
  7 questions. Likert scale: never; almost never; sometimes; fairly often; very often.
Severity of Acute Stress Symptoms | one-week (post)
  7 questions. Likert scale: never; almost never; sometimes; fairly often; very often.
Brief Resilience Scale | baseline (pre)
  6 questions. Likert scale: strongly disagree; disagree; neutral; agree; strongly agree
Brief Resilience Scale | one-week (post)
  6 questions. Likert scale: strongly disagree; disagree; neutral; agree; strongly agree
Daily Stress Scale | baseline (pre)
  6 questions. Numeric rating scale from 0-10. O indicating no stress and 10 indicating extremly stressful.
Daily Stress Scale | one-week (post)
  6 questions. Numeric rating scale from 0-10. O indicating no stress and 10 indicating extremly stressful.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sullivan, DC, PhD, Study Director — Life University Center for Chiropractic Research
Locations (1):
- Life University Center for Chiropractic Research, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No